CLINICAL TRIAL: NCT02431013
Title: A Randomized, Open-label, Multiple-dose, Parallel Study to Investigate The Effect of Cilostazol on the Disposition of Simvastatin in Healthy Male Volunteers
Brief Title: Cilostazol-Simvastatin Drug Interaction Study
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ajou University School of Medicine (Other)
Responsible Party: Principal Investigator, Doo-Yeoun Cho, Assistant Professor, Ajou University School of Medicine
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: DDI-103
Record Dates: First submitted 2015-04-23; First posted 2015-04-30 (Estimated); Last update posted 2015-05-01 (Estimated); Status verified 2015-04

CONDITIONS: Dyslipidemias; Peripheral Artery Disease
Keywords: Drug-drug interaction; Pharmacokinetics
MeSH Terms: conditions — Dyslipidemias; Peripheral Arterial Disease | interventions — Simvastatin; Pravastatin; Cilostazol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Simvastatin+Cilostazol (Experimental): Simvastatin 40 mg on Day 1. Cilostazol 100 mg twice a day for 6 days. Simvastatin 40 mg and Cilostazol 100 mg twice a day on Day 8.
  Interventions: Drug: Simvastatin; Drug: Cilostazol
- Pravastatin+Cilostazol (Active Comparator): Pravastatin 20 mg on Day 1. Cilostazol 100 mg twice a day for 6 days. Pravastatin 20 mg and Cilostazol 100 mg twice a day on Day 8.
  Interventions: Drug: Pravastatin; Drug: Cilostazol

INTERVENTIONS:
Drug: Simvastatin — Simvastatin 40 mg on Day 1 & Day 8.
  Other Names: S
  Arms: Simvastatin+Cilostazol
Drug: Pravastatin — Pravastatin 20 mg on Day 1 & Day 8.
  Other Names: P
  Arms: Pravastatin+Cilostazol
Drug: Cilostazol — Cilostazol 100 mg twice a day for 6 days & on Day 8 with statin.
  Other Names: C

SUMMARY:
This is a randomized, open-label, single & multiple-dose, parallel study to investigate the effect of cilostazol on the disposition of simvastatin & pravastatin in healthy male volunteers

DETAILED DESCRIPTION:
Eligibility for participation of this study will be determined from demographic information, medical history, physical examination, electrocardiogram (ECG) and clinical laboratory tests within 4 weeks before study drug administration. Subjects suitable for this study will be admitted to the Clinical Trial Center of Ajou University Medical Center on the day before dosing (Day -1).

On Day 1, Subjects will be dosed simvastatin 40 mg or pravastatin 20 mg. Pharmacokinetic samplings and blood pressure/pulse rate measurement will be done upto 24 hours after dosing.

From Day 2 ~ 7, Subjects will be dosed cilostazol 100 mg twice a day. On Day 8, Subjects will be dosed simvastatin 40 mg or pravastatin 20 mg with cilostazol 100 mg twice a day. Pharmacokinetic samplings and blood pressure/pulse rate measurement will be done upto 24 hours after dosing.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male subjects aged 20 - 45 years
* With in 20% of ideal body weight, {Ideal body weight=[height(cm)-100]*0.9}
* Agreement with written informed consent

Exclusion Criteria:

* Clinically significant cardiovascular, pulmonary, hepatic, renal, hematologic, gastrointestinal disease or mental disorder (Past history or present)
* Inadequate result of laboratory test (especially, AST/ALT > 1.25 x UNL, Total bilirubin > 1.5 x UNL)
* Positive reaction in the HBs Ag, anti-HCV Ab, anti-HIV Ab, VDRL test
* Taking OTC(Over the counter)medicine including oriental medicine within 7 days
* Clinically significant allergic disease (Except for mild allergic rhinitis and dermatitis seems to be not need for medication)
* Subject with known for hypersensitivity reaction to Cilostazol, Simvastatin or Pravastatin
* Previous whole blood donation within 60 days or component blood donation within 30 days
* Previous participation of other trial within 90 days
* Continued taking caffeine (caffeine > 5 cup/day), drinking (alcohol > 30 g/day) and severe heavy smoker (cigarette > 1/2 pack per day)
* An impossible one who participates in clinical trial by investigator's decision including for reason of laboratory test result

Ages: 20 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Estimated)
Dates: Start 2015-04; Primary Completion 2015-08 (Estimated)

PRIMARY OUTCOMES:
AUC (area under the time-concentration curve) of Simvastatin | up to 12 hours after Simvastatin dosing

SECONDARY OUTCOMES:
Cmax (maximum plasma concentration) of Simvastatin | up to 12 hours after Simvastatin dosing
Cmax (maximum plasma concentration) of Pravastatin | up to 12 hours after Pravastatin dosing
AUC (area under the time-concentration curve) of Pravastatin | up to 12 hours after Pravastatin dosing

CONTACTS AND LOCATIONS:
Overall Officials: Doo-Yeoun Cho, MD, Principal Investigator — Ajou University School of Medicine
Locations (1):
- Ajou University Medical Center, Suwon, Gyeonggi-do, South Korea